CLINICAL TRIAL: NCT03160807
Title: An Open Label Non Placebo Study to Evaluate Efficacy and Safety of Levofloxacin as an Empirical Therapy in Patients With Complicated Urinary Tract Infections
Brief Title: Levofloxacin as an Empirical Therapy in Patients With Complicated Urinary Tract Infections
Acronym: Levolet-KZ16
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EM_KZ_LEVOLET
Record Dates: First submitted 2016-06-28; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levofloxacin 5 days (Experimental): Levolet 500 mg given for 5 days
  Interventions: Drug: Levofloxacin
- Levofloxacin 10 days (Active Comparator): Levolet 500 mg given for 10 days
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin — Levolet 500 mg OD for 5 days
  Other Names: Levolet 500
  Arms: Levofloxacin 5 days
Drug: Levofloxacin — Levolet 500 OD for 10 days
  Other Names: Levolet 500
  Arms: Levofloxacin 10 days

SUMMARY:
Study is planned to evaluate safety and efficacy of Levolet in patients with complicated UTI

DETAILED DESCRIPTION:
A complicated urinary tract infection is a urinary infection occurring in a patient with a structural or functional abnormality of the genitourinary tract.

Fluoroquinolones have been recommended as the antimicrobials of choice for the empirical treatment of complicated urinary tract. Levofloxacin is a broad spectrum agent, which is known to demonstrate good clinical efficacy against urinary tract infection (UTI).

There is no published evidence available on the empirical use of Levofloxacin 500 mg OD and its optimal duration of therapy in patients with Complicated Urinary Tract Infections (cUTI). The present study evaluates the efficacy and safety, and optimal duration of therapy of levofloxacin 500 mg OD in patients with complicated UTI.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women over 18 years of age with cUTI in
* One or more clinical symptoms and signs of a lower UTI: fever (> 38°C, orally), chills, frequency of micturition, dysuria, urge sensation.
* One or more of the following underlying conditions suggestive of cUTI:
* Indwelling urinary catheter.
* Neurogenic bladder.
* Obstructive uropathy due to lithiasis, tumor or fibrosis.
* Acute urinary retention in men

Exclusion Criteria:

* History of allergy to quinolones
* Are unable to take oral medication
* Have an intractable infection requiring > 14 days of therapy
* Have a requirement for concomitant administration of sucralfate or divalent and trivalent cations such as iron or antacids containing magnesium, aluminum or calcium
* Have prostatitis or epididymitis
* Have had a renal transplant
* Have ileal loop or vesica- urethral reflux
* Have significant liver or kidney impairment
* Have a history of tendinopathy associated with fluoroquinolones
* Are pregnant, nursing
* Have a history of convulsions or CNS disorders

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with clinical cure rates at test of cure visit (TOC) defined as follows- Cure: a complete resolution of clinically significant signs & symptoms | Baseline to 5 days
  Cure: a complete resolution of clinically significant signs & symptoms

SECONDARY OUTCOMES:
Percentage of patients with microbiological eradication at test of cure visit (TOC) | Baseline to 5 days and upto 10 days
  Eradication: All uropathogens present at ≥105 CFU/ml at baseline had been reduced to <104 CFU/ml
No. of adverse events in entire study duration | Baseline to EOT visit (Baseline to 15 days)
  Type and total number of AEs recorded in study duration
Percentage of patient compliant to therapy in each study arm. | Baseline to EOT visit (Baseline to 15 days)
  Percentage of patients compliant to study treatment
Percentage of patient samples sensitive to levofloxacin in each study arm. | Baseline to EOT (Baseline to 15 days)
  Percent sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ilyas Tungiskhanovich, Principal Investigator — Scientific Centre of Urology named after B.U Dzharbusynov 2, Basenov street, Almaty 050060, Republic of Kazakhstan
Locations (1):
- Scientific Centre of Urology named after B.U Dzharbusynov 2, Basenov street,, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes